CLINICAL TRIAL: NCT07216001
Title: Role of Omega-DEK in Childhood Apraxia of Speech
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Claudia R. Morris (Other)
Responsible Party: Sponsor-Investigator, Claudia R. Morris, Professor, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00007888
Record Dates: First submitted 2025-10-10; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Childhood Apraxia of Speech; Verbal Apraxia; Autism
MeSH Terms: conditions — Apraxias; Autistic Disorder | interventions — Carnitine

STUDY DESIGN:
Intervention Model Description: This study has a 12-week open-label trial of Omega-DEK plus L-carnitine followed by an 8-week placebo-controlled discontinuation where participants are randomized to continue Omega-DEK or take a placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omega-DEK and L-carnitine for 12 Weeks Followed by Omega-DEK for 8 Weeks (Experimental): Children aged 3 to 6 years old with confirmed childhood apraxia of speech (CAS) receiving Omega-DEK and L-carnitine for the 12-week open-label trial, who are then randomized to continue to receive Omega-DEK for 8 additional weeks.
  Interventions: Drug: Omega-DEK; Drug: L-carnitine
- Omega-DEK and L-carnitine for 12 Weeks Followed by Placebo for 8 Weeks (Experimental): Children aged 3 to 6 years old with confirmed childhood apraxia of speech (CAS) receiving Omega-DEK and L-carnitine for the 12-week open-label trial, who are then randomized to receive a placebo to match Omega-DEK for 8 weeks.
  Interventions: Drug: Omega-DEK; Drug: L-carnitine; Drug: Placebo

INTERVENTIONS:
Drug: Omega-DEK — Participants take 2 capsules, twice daily (BID).
Drug: L-carnitine — Participants take 250 mg L-carnitine administered as a 2.5 mL oral solution twice daily (BID). L-carnitine is provided to participants only during the 12-week open-label trial.
  Other Names: Carnitor®
Drug: Placebo — A placebo of palm kernel oil to match Omega-DEK is provided. Participants take 2 capsules, twice daily (BID).
  Arms: Omega-DEK and L-carnitine for 12 Weeks Followed by Placebo for 8 Weeks

SUMMARY:
This is a 20-week study for children between 3 and 6 years old with confirmed childhood apraxia of speech (CAS). The study includes a 12-week open-label pilot feasibility study of an investigational drug (Omega-DEK) plus L-carnitine (Carnitor®), which is followed by an 8-week randomized, placebo-controlled discontinuation period among the same study participants.

DETAILED DESCRIPTION:
Verbal apraxia (VA) is a severe neurological motor planning speech disorder of unknown etiology. It is a devastating disorder that is insufficiently recognized by general pediatricians and often goes unaddressed and improperly treated during critical years of speech and language development. The high prevalence of this disorder excludes it as an "orphan" disease, although like autism, it may have met the definition over a decade ago. However, inadequate awareness of this condition among practitioners renders it a neglected disorder. Confusion around this condition is reflected by the vast number of terms used to define it, including Childhood Apraxia of Speech, Developmental Apraxia, Developmental Dyspraxia, Speech Apraxia, and Speech Dyspraxia to name a few.

Approximately half of children with autism spectrum disorders (ASD) have some degree of apraxia, although not all apraxic children are autistic. There is currently no recognized cure for VA, and it is thought to be a life-long condition. Standard treatment is extremely costly and involves intensive and frequent 1:1 speech therapy with a speech pathologist knowledgeable in VA. Typical response to therapy tends to be slow, and some children do not learn how to talk, thereby requiring alternate means of communication. Children with this disorder find it very difficult to correctly pronounce sounds, syllables, and words, despite intense effort. Intelligibility is poor, and some children remain completely speechless and require the use of augmentative communication devices, sign language and/or a picture exchange communication system.

Many children with VA present with a unique but homogeneous group of neurological symptoms that affect coordination, muscle tone and sensory issues in addition to expressive speech delay, suggesting a common underlying mechanism of disease. Vitamin E (vit E) deficiency causes a constellation of symptoms that overlap those of speech apraxia, limb dyspraxia, hypotonia and sensory integration dysfunction (including abnormalities in proprioception, vestibular sensation, and pain interpretation) that often occur in VA and ASD. Low bioavailability of vit E will create an environment within the cell membrane where vital polyunsaturated fatty acids (PUFAs) are vulnerable to lipid peroxidation and early destruction. This can lead to a functional PUFA deficiency and neurological sequelae that may be reversible through supplementation with PUFA/vit E. In addition, PUFA supplementation increases utilization of vit E in the body. These two supplements may have synergistic effects at higher doses.

An unexpected number of apraxic children have a carnitine deficiency, high antigliadin antibodies and carry a gluten-sensitivity major histocompatibility complex (HLA), suggesting abnormal fatty acid metabolism, increased oxidative stress and a potential link to gastrointestinal inflammation and gluten-sensitivity that creates a distinctive nutritional requirement in these children that may benefit from an investigational drug specifically formulated to targets unique deficiencies that contribute to VA. The researchers speculate that patients with gluten sensitivity or those carrying a celiac HLA with autism/VA may not have classic celiac disease, but perhaps a broader diagnosis of gluten-sensitivity associated with malabsorption and neurobehavioral consequences of nutritional deficiencies that needs consideration. The less sensitive celiac biomarker, antigliadin immunoglobulin G (IgG), frequently found in both ASD and VA may represent a biomarker that identifies an intervention-responder group. A recent double-blind randomized, placebo-controlled trial in irritable bowel syndrome concluded that a non-celiac gluten intolerance my exist, a concept in need of exploration in both ASD and VA.

In this study, children between 3 and 6 years old with confirmed childhood apraxia of speech (CAS) will take an investigational drug (Omega-DEK) plus L-carnitine (Carnitor®) for 12 weeks. This open-label period of the study is followed by an 8-week blinded trial where participants will be randomized to continue taking Omega-DEK or to take a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of childhood apraxia of speech/verbal apraxia by a qualified professional (SLP) based on established guidelines.
2. Male and female, age 36 months - 6 years (inclusive)
3. Ability to comprehend and use Standard American English

Exclusion Criteria:

1. Children unable to tolerate oral supplementation
2. Known allergy to fish oil, palm kernel oil or other ingredients in investigational drug
3. Medical or genetic condition that in the opinion of the PI/Co-Is may affect participation and compromise results (including significant receptive language delay, moderate-severe cognitive delay, complex medical history, hearing loss, cerebral palsy, history of traumatic brain injury or severe anoxic event, Down's syndrome).
4. Known seizure disorder or history of febrile seizures
5. History of cardiac dysrhythmia or abnormal ECG at baseline
6. A prothrombin time test with an international normalised ratio (PT/INR) >1.2.
7. Use of blood thinners, including chronic aspirin, chronic NSAIDS, warfarin etc.
8. A history of PUFA or vit E supplementation use within 3 months prior to enrollment in the study
9. On an elimination diet for < 3 months (gluten, casein, yeast free etc.) prior to enrollment, or planning to initiate a special diet during the study
10. Recent reintroduction of food items from elimination diet < 3 months
11. On any additional nutritional interventions/supplements < 3 months (i.e. high dose vitamins/minerals that exceed what would be found in a children's multivitamin supplement etc., probiotics)
12. Any new chronic medication < 3 months prior to enrollment (stable doses > 3 months allowed; medications for acute illness allowed including antipyretics, antibiotics, asthma medication)
13. Anticipated initiation of new chronic medication during study timeline including new attention-deficit/hyperactivity disorder (ADHD) medications, other behavior medications
14. Plans to try additional complementary interventions or diets during the study period
15. Planned surgery during or within 4 weeks after conclusion of trial

Ages: 36 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percent of Participants Retained in Study | Up to Week 20
  Feasibility of the intervention is assessed with the percentage of enrolled participants who complete the 20 week study. Successful retention is defined as >85% of enrolled participants completing the study.

SECONDARY OUTCOMES:
Percent of Participants With Complete Outcome Data | Up to Week 20
  Feasibility of the intervention is assessed with the percentage of participants who complete all surveys and study visits. Successful collection of outcome data is defined as >90% of participants completing study surveys and visits.
Change in Dynamic Evaluation of Motor Speech Skill (DEMSS) Score | Baseline, Week 12, Week 20
  The Dynamic Evaluation of Motor Speech Skill (DEMSS) is a validated tool specifically designed to identify the level of breakdown in a child's ability to speak so that treatment can be established, and improvement tracked. The DEMSS is comprised of 9 subtests with a total of 66 utterances which are associated with 171 items. Four subscores for overall articulatory accuracy of the word, vowel accuracy, prosodic accuracy, and consistency, are calculated. An overall score is calculated and ranges from 0 to 426, where lower scores suggest that CAS is present. Within a clinical setting, scores between 0 and 323 indicate CAS, scores between 323 and 373 indicate mild evidence of mild CAS, and scores of 373 to 426 indicate little or no evidence of CAS. Baseline scores are compared to scores at Week 12, for analysis of the open-label portion of the study, while Week 12 and Week 20 scores are compared for analysis of the randomized discontinuation portion of the study.
Mean Length of Utterances (MLU) | Baseline, Week 12, Week 20
  Mean length of utterance (MLU) is an assessment of expressive language measures the average number of morphemes per utterance. Morphemes are smallest language elements that make up linguistic expression. A spontaneous speech sample will be obtained and MLU is calculated as the number of morphemes in each utterance divided by the total number of utterances.
Clinical Global Impression for Improvement Scale (CGI-I) Score | Weeks 1, 4, 8, 12 (during the open-label portion of the study), weekly during Weeks 13-22 (during the randomized portion of the study)
  The CGI-I is a 7-point scale designed to measure overall improvement from baseline. The CGI-I is rated by an independent evaluator who is blind to treatment assignment during the randomized discontinuation phase. Scores range from 1 (Very Much Improved) to 4 (Unchanged) to 7 (Very Much Worse). Positive response to treatment (an improvement from baseline) is defined by a rating of Much Improved or Very Much Improved. Scores of 3 (minimally improved), 4 (no change) and 5 (minimally worse) indicate no change. Scores of 6 or 7 are considered as a worsening of symptoms from baseline (a negative response).

CONTACTS AND LOCATIONS:
Overall Officials: Claudia R Morris, MD, Principal Investigator — Emory University; Lawrence Scahill, MSN,PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Marcus Autism Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for study outcomes and demographics will be made available for sharing with other researchers.
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing following publication of the primary and secondary outcomes for this study.
Access Criteria: Researchers wanting to share data from this study will need to submit a proposal for their planned research to Dr. Morris at claudia.r.morris@emory.edu.